CLINICAL TRIAL: NCT07192302
Title: the Treatment Strategy of Partial Rotator Cuff Injury in Stiff Shoulders
Brief Title: Partial Rotator Cuff Injury Combined With Stiff Shoulder
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hebei Medical University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GJL20250831
Record Dates: First submitted 2025-08-31; First posted 2025-09-25 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-08

CONDITIONS: Rotator Cuff Tears of the Shoulder; Shoulder Adhesive Capsulitis; Shoulder Arthroscopy
MeSH Terms: conditions — Bursitis | interventions — Arthroscopy; Administration, Inhalation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Early Surgery) (Experimental): : Arthroscopic surgery within 6 weeks
  Interventions: Procedure: Arthroscopy
- Group B (Rehabilitation-First) (Sham Comparator): 6-month structured physical therapy program. Patients who do not achieve a pre-defined successful outcome at 6 months will then undergo delayed surgery.
  Interventions: Drug: Drugs administration

INTERVENTIONS:
Procedure: Arthroscopy — Early Surgical Intervention in Patients with Partial Rotator Cuff Tears and Concomitant Shoulder Stiffness.
  Arms: Group A (Early Surgery)
Drug: Drugs administration — Oral Medication for Conservative Management of Partial Rotator Cuff Tears with Concomitant Shoulder Stiffness.
  Arms: Group B (Rehabilitation-First)

SUMMARY:
A Randomized Controlled Trial Comparing Early Surgical Intervention Versus a Structured Rehabilitation Program with Delayed Surgery if Needed for Partial-Thickness Rotator Cuff Tears with Concomitant Shoulder Stiffness: The SPIRIT Trial (Surgery for Partial Tears with Immobility Randomized Intervention Trial)

DETAILED DESCRIPTION:
Objective: To compare the clinical and functional outcomes of early surgical intervention (arthroscopic debridement/repair and capsular release) versus an initial structured, supervised rehabilitation program with delayed surgery only for non-responders, in patients with PTRCT and shoulder stiffness.

Methods: This will be a single-center, prospective, randomized, controlled, parallel-group trial. patients will be randomized (1:1) to either:

Group A (Early Surgery): Arthroscopic surgery within 6 weeks of randomization.

Group B (Rehabilitation-First): A 6-month structured physical therapy program. Patients who do not achieve a pre-defined successful outcome at 6 months will then undergo delayed surgery.

Primary outcome will be the change in the American Shoulder and Elbow Surgeons (ASES) Standardized Shoulder Assessment Score from baseline to 12 months. Secondary outcomes include pain (VAS), range of motion (ROM), Constant-Murley Score, Single Assessment Numeric Evaluation (SANE), and rates of conversion to surgery. Outcomes will be assessed at baseline 6 months and 6 months after surgery.

Expected Outcomes: The investigators hypothesize that the early surgery group will demonstrate faster initial improvement in pain and function. However, the investigators anticipate that by 6 months, a significant proportion of the rehabilitation-first group will avoid surgery altogether and achieve non-inferior, if not equivalent, outcomes compared to the early surgery group.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years.
2. Symptomatic shoulder pain for >2 weeks.
3. MRI-confirmed partial-thickness rotator cuff tear (>50% tendon thickness or >5mm in length).
4. Concomitant shoulder stiffness, defined as passive range of motion loss of ≥25% in at least two planes (forward flexion, abduction, external rotation, or internal rotation) compared to the contralateral side.
5. Failure of a brief (≥2 weeks) trial of conservative care (e.g., oral NSAIDs).

Exclusion Criteria:

1. Age< 18 or >80 years.
2. Full-thickness rotator cuff tear.
3. Previous surgery on the affected shoulder.
4. Glenohumeral osteoarthritis (Grade ≥2 Samilson-Prieto).
5. Cervical radiculopathy as a primary cause of symptoms.
6. Systemic inflammatory arthritis.
7. Neurologic disorder affecting the shoulder.
8. Contraindications to surgery or general anesthesia.
9. Inability to comply with the rehabilitation protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index （SPADI） | 6 month before surgery and 6 months after surgery
  Shoulder Pain and Disability Index （SPADI） from 0-100. The lower the number, the better the functional outcomes of the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Jialiang Guo, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No